CLINICAL TRIAL: NCT06739876
Title: Effects of a Wearable Device and Social Media-Based Intervention on Physical Activity and Sleep Quality in Adults: a Randomized Controlled Trial
Brief Title: Effects of a Wearable Device and Social Media-Based Intervention on Physical Activity and Sleep Quality in Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Chung Hsing University (Other)
Responsible Party: Principal Investigator, Po-Wen Ku, PhD, Professor, National Chung Hsing University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NCUEREC-110-082; 111-2410-H-005-055-MY3 (Other: National Science and Technology Council)
Record Dates: First submitted 2024-12-12; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Sleep; Physical Activity
Keywords: Sleep quality; wearable device; motivation; social media support; physical activity
MeSH Terms: conditions — Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants in the intervention group will wear a device and will either receive motivational support via social media or not. The control group will not wear a device during the intervention phase.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No wearable device: Control (No Intervention): The control group will not wear the device at times other than completing assessments at baseline, post-intervention, and follow-up.
- Intervention: Device and motivational support via social media (Experimental): Participants in the Device and motivational support group will wear the device (Garmin tracker) for a month. In addition, they will receive motivational support via social media.
  Interventions: Behavioral: Wearable device-based intervention (with motivational support via social media)
- Intervention: Device (Experimental): Participants in the Device group will wear the device (Garmin tracker) for a month.
  Interventions: Behavioral: Wearable device-based intervention (without support)

INTERVENTIONS:
Behavioral: Wearable device-based intervention (with motivational support via social media) — The wearable device-based intervention aims to reduce sedentary behavior as the Move alert function may facilitate the management of one's physical activity. Motivational support will be provided via an online community created using LINE platform. The platform serve for the following purposes: a) providing psychoeduation prior to the intervention; b) providing a place for participants to motivate and encourage each other; c) provide health knowledge to participants weekly, to motivate behavioral change; d) encouraging participants to upload their daily step count to the community page to motivate each other's progress; e) based on participant's performance, research assistants will provide tailored support using Line stickers designed for the present intervention; f) research assistants will monitor participants' step counts and provide prizes (vouchers) for those who had the most step counts and made the most improvements.
  Arms: Intervention: Device and motivational support via social media
Behavioral: Wearable device-based intervention (without support) — The wearable device-based intervention aims to reduce sedentary behavior as the Move alert function may facilitate the management of one's physical activity.
  Arms: Intervention: Device

SUMMARY:
The goal of this randomized controlled trial is to examine whether the use of a wearable device and social media based intention increases physical activity and enhance sleep quality among adults.

DETAILED DESCRIPTION:
The present study aims to study sedentary breaks and sleep quality in Taiwanese adults.

This is a three-arm randomized controlled trial, exploring the effects of a one-month wearable device-based intervention (Garmin tracker) in increasing physical activity and improving sleep quality in adults (Target n = 75 ). The one-month follow-up assessment will be conducted to examine the remaining effects of the intervention.

The main questions it aims to answer are:

Does using a wearable device improve physical activity and improve sleep quality among adults?

Does the inclusion of motivational support provided via social media promote even greater effects in increasing physical activity and improvements in sleep quality?

Researchers will compare groups wearing a device and receiving motivational support via social media (intervention group 1) or wearing a device but without support (intervention 2) to a control condition (participants who do not wear a device and do not receive support) to see whether a wearable device could increase physical activity and improve sleep.

ELIGIBILITY:
Inclusion Criteria:

* Those who have not used a wearable-device before.

Exclusion Criteria:

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity | Baseline, and post-assessment (immediately after the intervention), one month follow-up
  Change in physical activity will be assessed by self-report measure on sedentary breaks and behaviour (the measure was developed by the investigator in a previous study). In addition, it will also be assessed by a measurable device (physical activity-related parameters assessed by Garmin monitor).

SECONDARY OUTCOMES:
Change in sleep | Baseline, and post-assessment (immediately after the intervention), one month follow-up
  Description: Sleep will be assessed using the translated Athens Insomnia Scale. The total score will be used, ranging from 0 to 15. Higher scores indicate higher levels of insomnia problems. Objective sleep will also be assessed by a measurable device (via Garmin monitors).

OTHER OUTCOMES:
Satisfaction with life | Time Frame: Baseline, and post-assessment (immediately after the intervention), one month follow-up
  Satisfaction with life will be measured by the Satisfaction With Life Scale. The total score will be used, ranging from the minimum value of 5 to the maximum value of 35. Higher scores indicate higher satisfaction.
Stress | Time Frame: Baseline, and post-assessment (immediately after the intervention), one month follow-up
  Stress will be measured by the Perceived Stress Scale. The total score will be used, ranging from the minimum value of 0 to 56. A score of 0-28 indicate normal perceived stress levels, 29-42 indicate relatively high stress; a score of43-56 indicate high perceived stress. Greater values indicate greater levels of stress.
Depressive symptoms | Time Frame: Baseline, and post-assessment (immediately after the intervention), one month follow-up
  Depressive symptoms will be measured by the Center for Epidemiologic Studies Depression Scale. The total score will be used, ranging from the minimum value of 0 to the maximum value of 30. A score of 10 or above indicate depressive symptoms. Higher scores indicate higher levels of depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- National Chung Hsing University, Taichung, Taiwan